CLINICAL TRIAL: NCT03228394
Title: A Phase 2A, Double-blind, Placebo-controlled, Multiple-dose Escalation Study to Evaluate Safety, Pharmacokinetics and Efficacy of Intravenously Administered Ganaxolone in Women With Postpartum Depression
Brief Title: A Clinical Trial of Intravenous (IV) Ganaxolone in Women With Postpartum Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-PPD-2002
Record Dates: First submitted 2017-07-05; First posted 2017-07-24 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Depression; Depressive Disorder; Depression, Postpartum; Behavioral Symptoms; Mood Disorders; Mental Disorders; Puerperal Disorders; Pregnancy Complications; Postpartum; PPD
Keywords: Postpartum Care; Postpartum Depression
MeSH Terms: conditions — Depression; Depressive Disorder; Depression, Postpartum; Behavioral Symptoms; Mood Disorders; Mental Disorders; Puerperal Disorders; Pregnancy Complications | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ganaxolone (Experimental): Intravenous
  Interventions: Drug: Ganaxolone
- Placebo (Placebo Comparator): Intravenous
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ganaxolone — Ganaxolone IV
  Arms: Ganaxolone
Drug: Placebo — Placebo IV
  Arms: Placebo

SUMMARY:
This study will evaluate the Safety, Pharmacokinetics and Efficacy of IV Administration of Ganaxolone in Women with Postpartum Depression

DETAILED DESCRIPTION:
This study will explore whether ganaxolone is safe and well tolerated in women suffering from PPD. In addition, ganaxolone's efficacy in treating depressive symptoms will be assessed through a set of exploratory analyses. Plasma levels of ganaxolone will be determined through pharmacokinetic analysis. The study results will be used to select a ganaxolone dose and dosing regimen for further development in PPD.

ELIGIBILITY:
Inclusion Criteria:

* Participant experienced a Major Depressive Episode, which started between the start of the third trimester and 4 weeks following delivery. The Major Depressive Episode must be diagnosed according to Mini International Neuropsychiatric Interview (MINI) 7.0 interview
* Participant gave birth in the last 6 months
* Participant has a Hamilton Depression Rating Scale 17-item version (HAMD17) score of ≥ 26 at screening
* Participant must agree to stop breastfeeding from start of study treatment or must agree to temporarily cease giving breast milk to her infant(s)

Exclusion Criteria:

* Current or past history of any psychotic illness, including Major Depressive Episode with psychotic features
* History of suicide attempt within the past 3 years
* Active suicidal ideation
* History of bipolar I disorder
* History of seizure disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with postpartum depression
Enrollment: 91 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2020-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Marinus Research Site, Little Rock, Arkansas
  - Marinus Research Site, Costa Mesa, California
  - Marinus Research Site, Lemon Grove, California
  - Marinus Research Site, San Diego, California
  - Marinus Research Site, Jacksonville, Florida
  - Marinus Research Site, Atlanta, Georgia
  - Marinus Research Site, Decatur, Georgia
  - Marinus Research Site, Leawood, Kansas
  - Marinus Research Site, Overland Park, Kansas
  - Marinus Research Site, New York, New York
  - Marinus Research Site, Dayton, Ohio
  - Marinus Research Site, Houston, Texas
  - Marinus Research Site, Irving, Texas
  - Marinus Research Site, Orem, Utah
  - Marinus Research Site, Salt Lake City, Utah
  - Marinus Research Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Cohort 1: Intravenous (IV) infusion of placebo (PBO) at rate of 16 milliliter per hour (mL/h) for 48 hours, then 8 mL/h for 12 hours
- Ganaxolone Cohort 1: IV infusion of ganaxolone (GNX) at rate of 4 milligram per hour (mg/h) (16 mL/h) for 48 hours, then 2 mg/h for 12 hours
- Placebo Cohort 2: IV infusion of PBO at rate of 16 mL/h for 48 hours, then 8 mL/h for 12 hours.
- Ganaxolone Cohort 2: IV infusion of GNX at rate of 8 mg/h for 48 hours, then 4 mg/h (8 mL/h) for 12 hours
- Placebo Cohort 3: IV bolus of 24 mL PBO over 2 minutes; then 24 mL for 48 hours and then 12 mL/h for 12 hours.
- Ganaxolone Cohort 3: IV bolus of 12 mg (24mL) GNX over 2 minutes; then GNX at 12 mg/h (24 mL/h) for 48 hours and then 6 mg/h (12 mL/h) for 12 hours.
- Placebo Cohort 6: IV infusion of PBO at rate of 40 mL/h for 6 hours; then 900 mg PBO (4 capsules) orally at dinner for 28 days
- Ganaxolone Cohort 6: IV infusion of GNX at rate of 20 mg/h (40 mL/h) for 6 hours followed by 900 mg (4 capsules) orally at dinner for 28 days
Period: Overall Study
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Started | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16
Completed | 4 | 5 | 12 | 13 | 10 | 10 | 12 | 13
Not Completed | 0 | 0 | 2 | 2 | 0 | 0 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Cohort 1; Placebo Cohort 2: IV infusion of PBO at rate of 16 mL/h for 48 hours, then 8 mL/h for 12 hours
- Ganaxolone Cohort 1: IV infusion of GNX at rate of 4 mg/h (16 mL/h) for 48 hours, then 2 mg/h for 12 hours
- Placebo Cohort 3: IV bolus of 24 mL PBO over 2 minutes; then 24 mL/h for 48 hours and then 12 mL/h for 12 hours
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6 | Total
Number analyzed (Participants) | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (2.22) | 24.4 (6.27) | 26.4 (6.02) | 27.0 (7.11) | 26.4 (5.70) | 25.0 (4.11) | 24.9 (5.10) | 28.8 (4.97) | 26.30 (3.495)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16 | 91
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 7
  Not Hispanic or Latino | 2 | 4 | 14 | 14 | 10 | 9 | 17 | 14 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 2 | 8 | 10 | 7 | 8 | 12 | 8 | 56
  White | 3 | 3 | 5 | 4 | 2 | 1 | 4 | 8 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale 17-item Version (HAMD17) Total Score
Description: The HAMD17 was a 17-item clinician-rated instrument used to assess the range of symptoms that were most frequently observed in participants with major depression. All items were scored on an ordinal scale between 0 and 4 (8 items) or 0 and 2 (9 items) of increasing severity. Each of 17 items was rated by clinician with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items, where 0 indicated no depression and 52 indicated severe depression. Higher score represented more severe condition. Baseline was defined as the Day 1 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and Day 3 post-infusion (60 hours post start of infusion) for Cohorts 1 to 3 and Baseline and Day 29 for Cohort 6
Population: Modified intent-to-treat (mITT) population: Included all participants in the safety set who had ≥1 post-randomization efficacy assessment. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 9 | 14 | 15
Scores on a scale
  Day 3 post-infusion (60 hours post start of infusion): number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 9 | 0 | 0
  Day 3 post-infusion (60 hours post start of infusion) | -13.0 (10.10) | -12.0 (6.82) | -14.0 (9.10) | -14.3 (10.23) | -11.0 (6.58) | -11.3 (7.04) |  |
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  Day 29 |  |  |  |  |  |  | -13.6 (11.51) | -11.5 (11.43)

2. Secondary Outcome: Change From Baseline in HAMD17 Total Score at Indicated Time Points
Description: as for outcome 1
Time Frame: Baseline, Day1 post-infusion(6hours post start of infusion), Day1(12hours post start of infusion), Day2(24hours post start of infusion),Day3 post-infusion(48hours post start of infusion),Day4(72hours post start of infusion),Days 8,11,15,22,36,57 and 71
Population: mITT population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Number analyzed (Participants) | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16
Scores on a scale
  Day 1 post-infusion (6 hours post start of infusion): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 16
  Day 1 post-infusion (6 hours post start of infusion) |  |  |  |  |  |  | -3.2 (6.85) | -6.1 (9.97)
  Day 1 (12 hours post start of infusion): number analyzed (Participants) | 4 | 5 | 13 | 11 | 10 | 8 | 0 | 0
  Day 1 (12 hours post start of infusion) | -3.8 (7.18) | -2.4 (1.52) | -3.2 (6.44) | -2.7 (5.59) | -1.9 (4.20) | 0.3 (2.92) |  |
  Day 2 (24 hours post start of infusion): number analyzed (Participants) | 4 | 5 | 14 | 14 | 10 | 9 | 17 | 16
  Day 2 (24 hours post start of infusion) | -8.0 (9.80) | -3.8 (5.31) | -6.4 (7.33) | -10.1 (8.90) | -5.2 (7.89) | -3.4 (4.13) | -5.1 (5.07) | -7.8 (8.07)
  Day 3 post-infusion (48 hours post start of infusion): number analyzed (Participants) | 4 | 5 | 13 | 14 | 10 | 10 | 0 | 0
  Day 3 post-infusion (48 hours post start of infusion) | -10.8 (12.09) | -11.0 (3.67) | -10.5 (9.26) | -13.7 (11.68) | -8.7 (7.15) | -11.2 (4.98) |  |
  Day 4 (72 hours post start of infusion): number analyzed (Participants) | 4 | 5 | 13 | 15 | 10 | 10 | 16 | 13
  Day 4 (72 hours post start of infusion) | -12.8 (14.73) | -10.2 (10.06) | -14.5 (9.12) | -17.3 (9.22) | -14.0 (6.72) | -10.5 (8.57) | -7.8 (6.83) | -7.0 (6.16)
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  Day 8 |  |  |  |  |  |  | -8.7 (8.99) | -8.7 (9.17)
  Day 11: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 9 | 11 | 11
  Day 11 | -13.3 (11.79) | -6.2 (5.72) | -9.7 (9.67) | -14.0 (12.56) | -8.2 (7.80) | -8.9 (9.65) | -13.6 (7.58) | -13.6 (9.84)
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 13
  Day 15 |  |  |  |  |  |  | -11.6 (8.38) | -12.7 (9.72)
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Day 22 |  |  |  |  |  |  | -12.3 (10.50) | -12.7 (9.55)
  Day 36: number analyzed (Participants) | 4 | 5 | 11 | 12 | 10 | 9 | 12 | 15
  Day 36 | -17.0 (12.46) | -11.0 (9.62) | -13.3 (6.48) | -16.5 (10.10) | -9.1 (8.70) | -11.1 (12.25) | -13.5 (10.76) | -13.0 (10.11)
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
  Day 57 |  |  |  |  |  |  | -16.0 (9.70) | -12.0 (9.49)
  Day 71: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 13
  Day 71 |  |  |  |  |  |  | -19.0 (7.87) | -14.8 (11.52)

3. Secondary Outcome: Number of Participants With HAMD17 Response
Description: HAMD17 Response was defined as ≥50% reduction from Baseline in total score. The HAMD17 was a 17-item clinician-rated instrument used to assess the range of symptoms that were most frequently observed in participants with major depression. All items were scored on an ordinal scale between 0 and 4 (8 items) or 0 and 2 (9 items) of increasing severity. Each of 17 items was rated by clinician with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items, where 0 indicated no depression and 52 indicated severe depression. Higher score represented more severe condition. Number of participants with HAMD17 response is presented.
Time Frame: Day1 post-infusion (6 hours post start of infusion [SOI]), Day 1 (12 hours post SOI), Day 2 (24 hours post SOI),Day 3 post-infusion (48 hours post SOI), Day 3 post-infusion (60 hours post SOI), Day 4 (72 hours post SOI), Days 8,11,15,22,29,36,57 and 71
Population: mITT population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Ganaxolone Cohort 3: IV bolus of GNX 12 mg (24mL) over 2 min; then 12 mg/h (24mL/h) for 48hrs.
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Number analyzed (Participants) | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16
Participants
  Day 1 post-infusion (6 hours post start of infusion): Responder: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 16
  Day 1 post-infusion (6 hours post start of infusion): Responder |  |  |  |  |  |  | 2 | 5
  Day 1 (12 hours post start of infusion): Responder: number analyzed (Participants) | 4 | 5 | 13 | 11 | 10 | 8 | 0 | 0
  Day 1 (12 hours post start of infusion): Responder | 0 | 0 | 1 | 0 | 0 | 0 |  |
  Day 2 (24 hours post start of infusion): Responder: number analyzed (Participants) | 4 | 5 | 14 | 14 | 10 | 9 | 17 | 16
  Day 2 (24 hours post start of infusion): Responder | 1 | 0 | 4 | 4 | 2 | 0 | 1 | 6
  Day 3 post-infusion (48 hours post start of infusion): Responder: number analyzed (Participants) | 4 | 5 | 13 | 14 | 10 | 10 | 0 | 0
  Day 3 post-infusion (48 hours post start of infusion): Responder | 2 | 1 | 6 | 7 | 4 | 4 |  |
  Day 3 post-infusion (60 hours post start of infusion): Responder: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 9 | 0 | 0
  Day 3 post-infusion (60 hours post start of infusion): Responder | 2 | 2 | 7 | 7 | 3 | 5 |  |
  Day 4 (72 hours post start of infusion): Responder: number analyzed (Participants) | 4 | 5 | 13 | 15 | 10 | 10 | 16 | 13
  Day 4 (72 hours post start of infusion): Responder | 2 | 3 | 7 | 11 | 6 | 5 | 3 | 3
  Day 8: Responder: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  Day 8: Responder |  |  |  |  |  |  | 4 | 5
  Day 11: Responder: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 9 | 11 | 11
  Day 11: Responder | 2 | 1 | 5 | 5 | 3 | 3 | 6 | 6
  Day 15: Responder: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 13
  Day 15: Responder |  |  |  |  |  |  | 8 | 6
  Day 22: Responder: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Day 22: Responder |  |  |  |  |  |  | 7 | 8
  Day 29: Responder: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  Day 29: Responder |  |  |  |  |  |  | 8 | 7
  Day 36: Responder: number analyzed (Participants) | 4 | 5 | 11 | 12 | 10 | 9 | 12 | 15
  Day 36: Responder | 3 | 3 | 5 | 7 | 4 | 5 | 6 | 8
  Day 57: Responder: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
  Day 57: Responder |  |  |  |  |  |  | 8 | 6
  Day 71: Responder: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 13
  Day 71: Responder |  |  |  |  |  |  | 9 | 9

4. Secondary Outcome: Number of Participants With HAMD17 Remission
Description: HAMD17 Remission was defined as total score ≤7. The HAMD17 was a 17-item clinician-rated instrument used to assess the range of symptoms that were most frequently observed in participants with major depression. All items were scored on an ordinal scale between 0 and 4 (8 items) or 0 and 2 (9 items) of increasing severity. Each of 17 items was rated by clinician with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items, where 0 indicated no depression and 52 indicated severe depression. Higher score represented more severe condition. Number of participants with HAMD17 remission is presented
Time Frame: Day1 post-infusion (6 hours post start of infusion [SOI]), Day 1 (12 hours post SOI), Day2 (24 hours post SOI), Day 3 post-infusion (48 hours post SOI), Day 3 post-infusion (60 hours post SOI), Day 4 (72 hours post SOI), Days 8,11,15,22,29,34,57 and 71
Population: mITT population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Number analyzed (Participants) | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16
Participants
  Day 1 post-infusion (6 hours post start of infusion): Remission: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 16
  Day 1 post-infusion (6 hours post start of infusion): Remission |  |  |  |  |  |  | 0 | 3
  Day 1 (12 hours post start of infusion): Remission: number analyzed (Participants) | 4 | 5 | 13 | 11 | 10 | 8 | 0 | 0
  Day 1 (12 hours post start of infusion): Remission | 0 | 0 | 0 | 0 | 0 | 0 |  |
  Day 2 (24 hours post start of infusion): Remission: number analyzed (Participants) | 4 | 5 | 14 | 14 | 10 | 9 | 17 | 16
  Day 2 (24 hours post start of infusion): Remission | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Day 3 post-infusion (48 hours post start of infusion): Remission: number analyzed (Participants) | 4 | 5 | 13 | 14 | 10 | 10 | 0 | 0
  Day 3 post-infusion (48 hours post start of infusion): Remission | 1 | 0 | 3 | 3 | 1 | 2 |  |
  Day 3 post-infusion (60 hours post start of infusion): Remission: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 9 | 0 | 0
  Day 3 post-infusion (60 hours post start of infusion): Remission | 1 | 1 | 4 | 4 | 2 | 2 |  |
  Day 4 (72 hours post start of infusion): Remission: number analyzed (Participants) | 4 | 5 | 13 | 15 | 10 | 10 | 16 | 13
  Day 4 (72 hours post start of infusion): Remission | 2 | 1 | 4 | 7 | 3 | 3 | 2 | 0
  Day 8: Remission: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  Day 8: Remission |  |  |  |  |  |  | 2 | 3
  Day 11: Remission: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 9 | 11 | 11
  Day 11: Remission | 1 | 0 | 3 | 5 | 2 | 1 | 4 | 3
  Day 15: Remission: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 13
  Day 15: Remission |  |  |  |  |  |  | 4 | 3
  Day 22: Remission: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Day 22: Remission |  |  |  |  |  |  | 4 | 5
  Day 29: Remission: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  Day 29: Remission |  |  |  |  |  |  | 6 | 4
  Day 34: Remission: number analyzed (Participants) | 4 | 5 | 11 | 12 | 10 | 9 | 12 | 15
  Day 34: Remission | 3 | 1 | 4 | 5 | 2 | 4 | 5 | 4
  Day 57: Remission: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
  Day 57: Remission |  |  |  |  |  |  | 6 | 4
  Day 71: Remission: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 13
  Day 71: Remission |  |  |  |  |  |  | 7 | 6

5. Secondary Outcome: Change From Baseline in Edinburgh Postnatal Depression Scale (EPDS) Total Score
Description: The EPDS is a validated 10-question depression assessment for postpartum women, which includes anxiety symptoms and excludes constitutional symptoms associated with depression common in the postpartum period, such as changes in sleeping patterns. It consists of 10 multiple choice questions with scores for each question ranging from 0-3. Questions 1, 2, & 4 are scored 0, 1, 2 or 3 with top box scored as 0 and the bottom box scored as 3. Questions 3 and 5 to 10 are reverse scored, with the top box scored as a 3 and the bottom box scored as 0. Scores are then summed for a total score, which ranges from 0: no depression to 30: severe depression. Higher score indicates severe depression. Baseline was defined as the Day 1 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline, Day 1, Day 2, Day 3 post-infusion (60 hours post start of infusion), Day 8, Day 11, Day 15, Day 22, Day 29, Day 34, Day 36, Day 57 and Day 71
Population: mITT population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Number analyzed (Participants) | 4 | 5 | 13 | 13 | 10 | 10 | 17 | 16
Scores on a scale
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 16
  Day 1 |  |  |  |  |  |  | -1.9 (2.87) | -5.4 (6.61)
  Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 16
  Day 2 |  |  |  |  |  |  | -4.9 (4.76) | -7.5 (5.81)
  Day 3 post-infusion (60 hours post start of infusion): number analyzed (Participants) | 4 | 5 | 13 | 13 | 10 | 10 | 0 | 0
  Day 3 post-infusion (60 hours post start of infusion) | -8.8 (14.64) | -8.0 (8.63) | -10.8 (6.66) | -10.8 (6.32) | -12.2 (6.21) | -10.9 (6.06) |  |
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 16
  Day 8 |  |  |  |  |  |  | -6.7 (6.01) | -9.6 (5.62)
  Day 11: number analyzed (Participants) | 4 | 5 | 12 | 13 | 10 | 10 | 0 | 0
  Day 11 | -13.5 (11.47) | -8.0 (4.12) | -9.6 (6.99) | -11.5 (8.02) | -8.8 (6.63) | -8.2 (7.35) |  |
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 15
  Day 15 |  |  |  |  |  |  | -8.0 (6.02) | -11.3 (5.06)
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  Day 22 |  |  |  |  |  |  | -8.2 (7.37) | -11.2 (6.13)
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 16
  Day 29 |  |  |  |  |  |  | -10.9 (8.14) | -10.0 (7.33)
  Day 34: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 10 | 0 | 0
  Day 34 | -14.5 (10.08) | -8.6 (5.32) | -9.8 (5.83) | -13.4 (5.81) | -9.1 (5.88) | -8.8 (8.27) |  |
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 14
  Day 36 |  |  |  |  |  |  | -11.8 (6.57) | -12.4 (6.57)
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
  Day 57 |  |  |  |  |  |  | -11.8 (6.79) | -9.4 (8.50)
  Day 71: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 13
  Day 71 |  |  |  |  |  |  | -14.0 (5.62) | -11.5 (7.34)

6. Secondary Outcome: Change From Baseline in Spielberger State-Trait Anxiety Inventory 6-item Version (STAI6) Total Score
Description: The STAI6 is a 6-item self-rated instrument used to assess anxiety state. The STAI6 questions included: 1. "I feel calm"; 2. "I am tense"; 3. "I feel upset"; 4. "I am relaxed"; 5. "I feel content"; 6. "I am worried". Each of these questions were rated as: a) "not at all"; b) "somewhat"; c) "moderately"; d) "very much". For questions 2, 3, and 6, the scoring was a = 1, b = 2, c = 3, and d = 4. For the other 3 questions, the scoring was a = 4, b = 3, c = 2, and d = 1. The STAI6 score was the result of first totaling the 6 individual item scores, and then prorating by a multiplication factor of 20/6 to acquire a score range of 20 (low anxiety) to 80 (high anxiety). Higher score indicated higher level of anxiety. Baseline was defined as the Day 1 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline, Day 1 (12 hours post start of infusion), Day 2, Day 3 post-infusion (60 hours post start of infusion), Day 4, Day 8, Day 11, Day 15, Day 22, Day 29, Day 34, Day 36, Day 57 and Day 71
Population: mITT population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Number analyzed (Participants) | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16
Scores on a scale
  Day 1 (12 hours post start of infusion): number analyzed (Participants) | 3 | 4 | 14 | 15 | 10 | 10 | 17 | 16
  Day 1 (12 hours post start of infusion) | -8.9 (20.09) | -4.2 (13.44) | -14.5 (14.48) | -12.01 (11.25) | -10.7 (10.52) | -11.3 (19.51) | -9.4 (14.78) | -17.7 (20.28)
  Day 2 | -9.2 (15.00) | -8.7 (13.25) | -15.0 (11.23) | -14.2 (17.88) | -12.7 (10.04) | -12.0 (13.07) | -12.9 (11.42) | -19.0 (17.96)
  Day 3 post-infusion (60 hours post start of infusion): number analyzed (Participants) | 4 | 5 | 13 | 13 | 10 | 10 | 0 | 0
  Day 3 post-infusion (60 hours post start of infusion) | -11.7 (33.39) | -22.0 (18.65) | -18.2 (12.95) | -21.0 (16.46) | -24.3 (16.11) | -24.0 (15.85) |  |
  Day 4: number analyzed (Participants) | 4 | 5 | 13 | 14 | 10 | 10 | 0 | 0
  Day 4 | -20.0 (23.73) | -20.7 (19.78) | -21.0 (13.77) | -22.9 (17.14) | -25.0 (13.99) | -22.3 (17.78) |  |
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 16
  Day 8 |  |  |  |  |  |  | -10.2 (18.88) | -15.6 (15.57)
  Day 11: number analyzed (Participants) | 4 | 5 | 12 | 13 | 10 | 10 | 0 | 0
  Day 11 | -21.7 (25.17) | -18.7 (20.22) | -16.9 (13.06) | -20.8 (17.17) | -17.0 (16.74) | -16.0 (15.93) |  |
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 14
  Day 15 |  |  |  |  |  |  | -12.3 (20.39) | -17.4 (19.00)
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 15
  Day 22 |  |  |  |  |  |  | -15.9 (15.88) | -21.8 (16.08)
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  Day 29 |  |  |  |  |  |  | -20.8 (13.89) | -18.9 (18.72)
  Day 34: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 10 | 0 | 0
  Day 34 | -20.8 (27.54) | -16.0 (21.53) | -16.1 (13.55) | -24.4 (13.80) | -18.7 (13.90) | -17.7 (20.37) |  |
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 14
  Day 36 |  |  |  |  |  |  | -21.9 (9.69) | -21.7 (19.07)
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
  Day 57 |  |  |  |  |  |  | -21.7 (12.67) | -13.3 (25.23)
  Day 71: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 13
  Day 71 |  |  |  |  |  |  | -31.7 (16.97) | -21.0 (16.91)

7. Secondary Outcome: Number of Participants With Response to Clinical Global Impression-Improvement (CGI-I) Scale
Description: The CGI-I scale is a clinician-rated 7-point scale used to assess how much the participant's illness had improved or worsened relative to a Baseline state at the beginning of the intervention. It was rated as: 1. "very much improved"; 2. "much improved"; 3. "minimally improved"; 4. "no change"; 5. "minimally worse"; 6. "much worse"; 7. "very much worse". Higher scores indicated worse condition. Response was defined as >50% decrease from Baseline in CGI-I total score.
Time Frame: Day 1 (12 hours post start of infusion), Day 2, Day 3 post-infusion (60 hours post start of infusion), Day 4, Day 8, Day 11, Day 15, Day 22, Day 29, Day 34, Day 36, Day 57 and Day 71
Population: mITT population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
Number analyzed (Participants) | 4 | 5 | 14 | 15 | 10 | 10 | 17 | 16
Participants
  Day 1 (12 hours post start of infusion): Very much or much improved | 0 | 0 | 2 | 3 | 1 | 0 | 3 | 7
  Day 1 (12 hours post start of infusion): Minimally or not improved | 4 | 5 | 12 | 12 | 9 | 10 | 14 | 9
  Day 2: Very much or much improved: number analyzed (Participants) | 4 | 5 | 13 | 15 | 10 | 10 | 17 | 16
  Day 2: Very much or much improved | 1 | 1 | 3 | 8 | 1 | 3 | 3 | 9
  Day 2: Minimally or not improved: number analyzed (Participants) | 4 | 5 | 13 | 15 | 10 | 10 | 17 | 16
  Day 2: Minimally or not improved | 3 | 4 | 10 | 7 | 9 | 7 | 14 | 7
  Day 3 post-infusion (60 hours post start of infusion): Very much or much improved: number analyzed (Participants) | 4 | 5 | 13 | 13 | 10 | 10 | 0 | 0
  Day 3 post-infusion (60 hours post start of infusion): Very much or much improved | 3 | 4 | 7 | 9 | 5 | 7 |  |
  Day 3 post-infusion (60 hours post start of infusion): Minimally or not improved: number analyzed (Participants) | 4 | 5 | 13 | 13 | 10 | 10 | 0 | 0
  Day 3 post-infusion (60 hours post start of infusion): Minimally or not improved | 1 | 1 | 6 | 4 | 5 | 3 |  |
  Day 4: Very much or much improved: number analyzed (Participants) | 4 | 5 | 13 | 15 | 10 | 10 | 0 | 0
  Day 4: Very much or much improved | 3 | 3 | 6 | 12 | 5 | 7 |  |
  Day 4: Minimally or not improved: number analyzed (Participants) | 4 | 5 | 13 | 15 | 10 | 10 | 0 | 0
  Day 4: Minimally or not improved | 1 | 2 | 7 | 3 | 5 | 3 |  |
  Day 8: Very much or much improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Day 8: Very much or much improved |  |  |  |  |  |  | 6 | 9
  Day 8: Minimally or not improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Day 8: Minimally or not improved |  |  |  |  |  |  | 9 | 6
  Day 11: Very much or much improved: number analyzed (Participants) | 4 | 5 | 12 | 13 | 10 | 10 | 0 | 0
  Day 11: Very much or much improved | 2 | 0 | 7 | 9 | 4 | 5 |  |
  Day 11: Minimally or not improved: number analyzed (Participants) | 4 | 5 | 12 | 13 | 10 | 10 | 0 | 0
  Day 11: Minimally or not improved | 2 | 5 | 5 | 4 | 6 | 5 |  |
  Day 15: Very much or much improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 15
  Day 15: Very much or much improved |  |  |  |  |  |  | 6 | 13
  Day 15: Minimally or not improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 15
  Day 15: Minimally or not improved |  |  |  |  |  |  | 10 | 2
  Day 22: Very much or much improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Day 22: Very much or much improved |  |  |  |  |  |  | 8 | 10
  Day 22: Minimally or not improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Day 22: Minimally or not improved |  |  |  |  |  |  | 7 | 5
  Day 29: Very much or much improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 16
  Day 29: Very much or much improved |  |  |  |  |  |  | 6 | 12
  Day 29: Minimally or not improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 16
  Day 29: Minimally or not improved |  |  |  |  |  |  | 10 | 4
  Day 34: Very much or much improved: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 10 | 0 | 0
  Day 34: Very much or much improved | 3 | 3 | 5 | 8 | 5 | 5 |  |
  Day 34: Minimally or not improved: number analyzed (Participants) | 4 | 5 | 12 | 12 | 10 | 10 | 0 | 0
  Day 34: Minimally or not improved | 1 | 2 | 7 | 4 | 5 | 5 |  |
  Day 36: Very much or much improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 14
  Day 36: Very much or much improved |  |  |  |  |  |  | 5 | 11
  Day 36: Minimally or not improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 14
  Day 36: Minimally or not improved |  |  |  |  |  |  | 7 | 3
  Day 57: Very much or much improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
  Day 57: Very much or much improved |  |  |  |  |  |  | 6 | 8
  Day 57: Minimally or not improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
  Day 57: Minimally or not improved |  |  |  |  |  |  | 6 | 4
  Day 71: Very much or much improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 13
  Day 71: Very much or much improved |  |  |  |  |  |  | 7 | 10
  Day 71: Minimally or not improved: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 13
  Day 71: Minimally or not improved |  |  |  |  |  |  | 5 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to 71 days
Arm/Group | Placebo Cohort 1 | Ganaxolone Cohort 1 | Placebo Cohort 2 | Ganaxolone Cohort 2 | Placebo Cohort 3 | Ganaxolone Cohort 3 | Placebo Cohort 6 | Ganaxolone Cohort 6
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/14 | 0/15 | 0/10 | 0/10 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/14 | 0/15 | 0/10 | 0/10 | 1/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/4 | 2/5 | 3/14 | 5/15 | 3/10 | 8/10 | 7/17 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Cohort 1 (N=4) | Ganaxolone Cohort 1 (N=5) | Placebo Cohort 2 (N=14) | Ganaxolone Cohort 2 (N=15) | Placebo Cohort 3 (N=10) | Ganaxolone Cohort 3 (N=10) | Placebo Cohort 6 (N=17) | Ganaxolone Cohort 6 (N=16)
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort 1 (N=4) | Ganaxolone Cohort 1 (N=5) | Placebo Cohort 2 (N=14) | Ganaxolone Cohort 2 (N=15) | Placebo Cohort 3 (N=10) | Ganaxolone Cohort 3 (N=10) | Placebo Cohort 6 (N=17) | Ganaxolone Cohort 6 (N=16)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling of Relaxation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coordination Abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 4 (8)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thinking Abnormal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eccymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Erythematous (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03228394/Prot_002.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT03228394/SAP_003.pdf